CLINICAL TRIAL: NCT02907372
Title: Impact of New Generation Hormono-therapy on Cognitive Functions in Elderly Patients Treated for a Metastatic Prostate Cancer
Acronym: COG-PRO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2016-001248-20
Record Dates: First submitted 2016-07-26; First posted 2016-09-20 (Estimated); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (CRPCa)
Keywords: cognitive dysfunctions; cognitive complaints; metastatic prostate cancer; new generations of hormone-therapy
MeSH Terms: conditions — Cognitive Dysfunction; Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- cognitive tests (Other)
  Interventions: Other: neuropsychologic evaluation; Other: oncogeriatric evaluation

INTERVENTIONS:
Other: neuropsychologic evaluation
Other: oncogeriatric evaluation

SUMMARY:
This study will assess the impact of the novel oral hormonal agents (abiraterone acetate or enzalutamide) among elderly metastatic prostate cancer patients. This study will assess the influence of treatments on patients' cognitive functions on a longitudinal basis and evaluate the quality of life and the adherence of patients who had or develop cognitive disorders.

DETAILED DESCRIPTION:
In this new area of multiples new treatments in advanced PCa that could be proposed to elderly patients, evaluating, understanding and analysing the incidence, severity of cognitive dysfunctions and their impact on quality of life, autonomy and adherence among this group of vulnerable patients with advanced disease is a challenge and is essential to help clinicians taking care of their patients. As the deficits may be subtle and not always related with complaints, cognitive functions need to be assessed by objective sensitive neuropsychological tests and by patient-perceived cognitive self-report questionnaire. In addition to the treatments,there is a range of potential confounders that can contribute to cognitive impairment, such as co-medications, psychological factors (e.g. anxiety or depression), fatigue, or cognitive reserve (i.e. patients with higher education, more occupational attainment, or participation in leisure activities report less clinical or cognitive changes with aging.

The evaluation and the comprehension of the cognitive decline in patients treated for a cancer are complex and need a multidisciplinary approach in human sciences in strong link to clinicians and biologist researchers.

Therefore, this study propose an original unique comprehensive interdisciplinary approach at the interface between public health, clinical research, psychology and biology which would have a direct impact on cancer patient care, including a consortium of neuropsychologists, oncologists and biologist researchers who are working together within the North West canceropole "cognition and cancer" program. In evaluating cognitive functions, mood, quality of life and adherence to treatments, fully in the scope of the proposal, will help to improve our knowledge in this new field of research in human health among cancer patients with a direct impact for the physicians and the patients. The strength of this project is to propose (in complement to the study conducted among patients) a comprehensive approach including an animal model with behavioural tasks as recommended by the ICCTF (International Cognition and Cancer Task Force).

This study will be the first one to address the question of the impact of the novel oral hormonal agents among elderly metastatic prostate cancer patients. This study will assess the influence of treatments on patients' cognitive functions on a longitudinal basis and evaluate the quality of life and the adherence of patients who had or develop cognitive disorders.

ELIGIBILITY:
Inclusion Criteria:

For the group of patients of interest :

* Patient must have a metastatic castration-resistant prostate cancer (CRPCa)
* Patient must be 70 years and more
* Performance Status 0-2
* Patient must have not received chemotherapy except one line per Docetaxel for hormono-sensitive situation and which must be completed for a least 18 months before inclusion
* Patient must have been already treated with first generation of androgen deprivation therapy
* Patient must be asymptomatic or pauci-symptomatic (with pain control, Visual Analog Scale ≤ 3)
* Patient must be candidate for a treatment by a new generation hormono-therapy (with abiraterone acetate or enzalutamide), in accordance to precautions of these treatments described in Summary Characteristics of Product and in combination with androgen deprivation therapy
* Treatment with biphosphonates is authorized
* No known brain metastasis
* Patient must be at least on level 3 on school scale
* Patient has signed informed consent

For the control group of patients :

* Patient with metastatic prostate cancer without resistance to castration
* Patient must be 70 years and more
* Performance Status 0-2
* Patient must have not received chemotherapy except one line per Docetaxel for hormono-sensitive situation and which must be completed for a least 18 months before inclusion
* Patient must have already started the first generation of androgen deprivation therapy at least since 3 months
* Patient must be asymptomatic or pauci-symptomatic (with pain control, Visual Analog Scale ≤ 3)
* No known brain metastasis
* Patient must be at least on level 3 on school scale
* Patient has signed informed consent

For the control group of healthy volunteers:

* Man
* No history of cancer,
* 70-year old or more,
* Health status consistent with the participation to the study
* At least on level 3 on school scale
* Signed informed consent

Exclusion Criteria:

For all participants (group of patients of interest, control group of patients and group of healthy volunteers):

* No previous treatment with a new generation hormone therapy (abiraterone acetate or enzalutamide)
* Neurological sequelae of (traumatic brain injury, stroke, multiple sclerosis, epilepsy, neuro-degenerative disease…)
* Known evolutive psychiatric disorder
* Drug use
* Heavy drinking
* Assessed to be unable or unwilling to comply with the requirements of the protocol

For group of patients of interest, additional non-inclusion criteria :

* Hypersensitivity to abiraterone acetate or enzalutamide
* For patients candidate for abiraterone acetate, presence of severe hepatic insufficiency

Min Age: 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 163 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
The proportion of elderly patients who will experience a decline in cognitive performances (at least for one cognitive function) by questionnaires | 3 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer

SECONDARY OUTCOMES:
The quantitative score of cognitive functions by questionnaires | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer
the quantitative score of quality of life by questionnaires for evaluate impact of cognitive impairment on quality of life to treatment | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer
the quantitative score of anxiety/depression by questionnaires for evaluate impact of cognitive impairment | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer
the quantitative score of fatigue by questionnaires for evaluate impact of cognitive impairment | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer
the quantitative score of autonomy by geriatric evaluation for evaluate impact of cognitive impairment | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer
the quantitative score of observance of treatment by questionnaire | Within 12 months after initiation of treatment by new generation hormono-therapies for a metastatic castration-resistant prostate cancer

CONTACTS AND LOCATIONS:
Locations (6):
- France (6):
  - CHU, Amiens
  - centre François Baclesse, Caen
  - Institut régional du Cancer de Montpellier (ICM), Montpellier
  - Chu Rouen, Rouen
  - Hôpital FOCH, Suresnes
  - IGR, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lange M, Laviec H, Castel H, Heutte N, Leconte A, Leger I, Giffard B, Capel A, Dubois M, Clarisse B, Coquan E, Di Fiore F, Gouerant S, Bartelemy P, Pierard L, Fizazi K, Joly F. Impact of new generation hormone-therapy on cognitive function in elderly patients treated for a metastatic prostate cancer: Cog-Pro trial protocol. BMC Cancer. 2017 Aug 16;17(1):549. doi: 10.1186/s12885-017-3534-8. PMID 28814281